CLINICAL TRIAL: NCT04560400
Title: Effects of Reading Direction and History of Multiple Concussions on King-Devick Test
Brief Title: Reverse King-Devick Test and History of Multiple Concussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1906713722
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No Concussion Conventional KD (Sham Comparator): Participants without concussion history perform conventional King-Devick Test.
  Interventions: Diagnostic Test: Conventional King-Devick test
- No Concussion Reverse KD (Active Comparator): Participants without concussion history perform reverse King-Devick Test.
  Interventions: Diagnostic Test: Reverse King-Devick test
- Single Concussion Conventional KD (Sham Comparator): Participants with 1 concussion history perform conventional King-Devick Test.
  Interventions: Diagnostic Test: Conventional King-Devick test
- Single Concussion Reverse KD (Active Comparator): Participants with 1 concussion history perform reverse King-Devick Test.
  Interventions: Diagnostic Test: Reverse King-Devick test
- Multiple Concussion Conventional KD (Sham Comparator): Participants with 2 or more concussion history perform conventional King-Devick Test.
  Interventions: Diagnostic Test: Conventional King-Devick test
- Multiple Concussion Reverse KD (Active Comparator): Participants with 2 or more concussion history perform reverse King-Devick Test.
  Interventions: Diagnostic Test: Reverse King-Devick test

INTERVENTIONS:
Diagnostic Test: Conventional King-Devick test — Conventional King-Devick test involves a series of number reading task from left to right and top to bottom, intending to test subjects' neuro-ophthalmologic function
  Arms: Multiple Concussion Conventional KD; No Concussion Conventional KD; Single Concussion Conventional KD
Diagnostic Test: Reverse King-Devick test — Reverse King-Devick test involves a series of number reading task from right to left and bottom to top, intending to test subjects' neuro-ophthalmologic function
  Arms: Multiple Concussion Reverse KD; No Concussion Reverse KD; Single Concussion Reverse KD

SUMMARY:
The purpose of this study is to examine the effects of concussion history and reading direction on baseline King- Devick Test (KDT) performance, a common component of sideline concussion assessments. The KDT is a timed assessment of saccades, or quick movements of the eyes between two points. This test is a form of rapid automatized naming and involved subjects reading digits arranged on a tablet screen as quickly and accurately as possible. The test has three progressively more challenging test "cards," as the horizontal guidelines between digits disappear from test card 1 to 2, and the vertical spacing between the lines of digits decreases from test card 2 to 3. KDT performance is evaluated in terms of both speed (duration to all three test cards) and the number of errors (digits read incorrectly or omitted). Previous studies have identified several factors that affect KDT performance aside from head injury, including age, sex, sleep deprivation, learning disabilities, and first languages other than English. History of concussion has not been shown to influence KDT performance. The investigators hypothesize that since the left-to-right (L-R) reading direction of the KDT is the same way in which to read English, the long-term effects of prior concussions on saccadic eye movements may be masked. The investigators want to answer the following three research questions: 1) What is the effect of KDT reading direction on baseline KDT performance? If the test is performed by reading digits in a right-to-left (R-L) direction, will KDT times be slower and the number of errors increase relative to a typical L-R KDT? 2) What is the effect of a history of multiple concussions on KDT performance relative to no history of concussion? 3) Is the R-L KDT more sensitive to a history of multiple concussions? The investigators hypothesize that individuals with a history of multiple concussions will perform significantly worse (longer test durations, more errors) than individuals with no concussion history on the R-L KDT. On the other hand, the investigators hypothesize that baseline performance on the traditional L-R KDT will not be able to discriminate individuals with a history of multiple concussions from those with no concussion history.

DETAILED DESCRIPTION:
Subjects will first be asked to complete a questionnaire. This questionnaire will collect demographic data (age, sex, years of education, native language and other languages spoken) and other pertinent data (vision correction, concussion history, ocular/visual injury and disorder history, learning disability diagnoses). The questionnaire will take approximately 3 minutes to complete.

Based on the concussion history provided in the questionnaire, the subject will be assigned to either Group NoHx (no concussion history) or Group HxMC (history of multiple concussions.) Then the subject will be randomized into one of two KDT formats: L-R KDT (natural reading direction) or R-L KDT (reverse reading direction) via a coin flip. The researcher will explain the KDT procedure by saying, "This test evaluates your saccadic eye movements, or rapid eye movements from one fixation point to the next. This test is comprised of three test cards. Each test card has eight lines of several digits (numbers). Please read the digits aloud as quickly but as accurately as possible from [L-R condition: 'left to right and top to bottom'; R-L condition: 'right to left and top to bottom']. If participants make a mistake, correct it if participants can and continue on. This is a timed test--tapping the tablet screen starts and stops the stopwatch. Participants will have a brief break in between cards to catch participants' breath. Each test card will get progressively harder. The horizontal lines guiding participants from digit to digit on each line on Test Card 1 disappear on Test Card 2. The lines of digits on Test Card 3 are closer together than they were on Test Card 2. Do you have any questions?"

The researcher will start the app and pull up the demonstration card for the L-R condition. For the R-L condition, the researcher will open a picture of the adapted demonstration card with the diagonal lines switched to indicate that subjects follow from the left-most digit to the right-most digit on the subsequent line. Subjects will complete the demonstration card twice according their condition instructions. Subjects will be reminded to "read the digits as quickly but accurately as possible" and in the direction according to their assigned test condition before starting the test. The researcher will silently count any errors while the subject completes each test card one at a time, taking a brief (1-2s) pause after tapping the screen to stop the timer and tapping again to start the timer and bringing up the next test card. At the conclusion of the test, the researcher will record the total time and number of errors on the subject data collection sheet. The subject will complete the test a second time, following the same instructions. The total time and number of errors for the second attempt will also be recorded. The investigators anticipate this portion of the data collection to take approximately 6 minutes. The total duration of the data collection will be approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 26 years old,
2. enrolled as an IU Bloomington student
3. a fluent English speaker.

Exclusion Criteria:

1. proficient fluency of any language that reads right to left (e.g. Arabic, Hebrew, Persian/ Farsi, Urdu Sindhi) or top to bottom and right to left (e.g. Japanese, Korean, or Chinese)
2. a history of only one diagnosed concussion
3. any visual, ocular, or brain injury within the past 12 months
4. any history of an eye movement disorder
5. any noncorrected visual impairment
6. a diagnosis of attention deficit/hyperactivity disorder, attention deficit disorder, dyslexia, dyscalculia, or a language processing disorder.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Between-group difference King-Devick test speed between conventional and reverse direction | Within 10 years of last concussion
  The comparison in King-Devick test speed (in second) between conventional reading direction of King-Devick test and reverse direction of King-Devick test will be made in each group (multiple concussion history, single concussion history, and no concussion history).
ROC diagnostic accuracy of reverse King-Devick test to differentiate concussion history | Within 10 years of last concussion
  ROC test will be performed to test the diagnostic accuracy of King-Devick test speed (in second), with reverse reading direction having superior diagnostic accuracy to identify individuals with multiple concussion history compared to the use of conventional reading direction of the King-Devick test.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided